CLINICAL TRIAL: NCT01433016
Title: Evaluation of the Capability of the ¹³C-Octanoate Breath Test (OBT) Measurement in Patients With Chronic Liver Disease to Differentiate Between Presence and Absence of HCC Determined by MRI
Brief Title: Detection of Hepatocellular Carcinoma (HCC) With Octanoate Breath ID Test Compared to MRI
Acronym: OBT for HCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to budgetary issues, the company has decided to focus on other applications at this stage.
Sponsor: Meridian Bioscience, Inc. (Industry)
Collaborators: Toronto General Hospital (Other); Medical University of South Carolina (Other); Northwestern University (Other); Henry Ford Health System (Other); Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCC-BID-0411
Record Dates: First submitted 2011-09-11; First posted 2011-09-13 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Chronic Liver Disease; Hepatocellular Carcinoma (HCC)
Keywords: HCC Hepatocellular carcinoma; OBT Octanoate Breath Test
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Octanaote Breath Test (Experimental): A Octanoate breath test will be performed on this single arm population
  Interventions: Drug: 13C Sodium Octanoate

INTERVENTIONS:
Drug: 13C Sodium Octanoate — 13C labeled Sodium Octanoate Substrate is provided in powder form in doses of 100mg for single breath test, and is dissolved in 150cc of tap water before ingestion. Duration of the observation after the drug ingestion is one hour.

SUMMARY:
The Exalenz clinical investigation is a multicenter, non-randomized, study of the ¹³C-Octanoate Breath Test (OBT). The present study is a feasibility trial, which aims to evaluate the capability of the OBT measurement to differentiate between presence and absence of HCC determined by Magnetic Resonance Imaging (MRI) in patients with chronic liver disease.

DETAILED DESCRIPTION:
The Octanoate Breath Test (OBT) developed by Exalenz is performed by the BreathID System consists of the BreathID device and a test kit containing a nasal cannula, a calibration gas container and a non-radioactive isotope ¹³C- Octanoate solution, and measures and computes the ratio between ¹³CO2 and 12CO2 in the patient's exhaled breath.

This study's aim is to provide data on this novel system to dynamically and accurately assess liver function at the bed side. It is hoped that the system will provide prognostic information faster than is achieved at present with traditional methods. It is hypothesized that in the future the OBT may have an impact on decision making and clinical practice in this group of HCC patients, allowing a greater chance for proper management and hence survival.

ELIGIBILITY:
Inclusion Criteria:

* Any patients with chronic liver disease at risk for HCC.
* Age > 18 years.
* Patient has an MRI result (positive or negative for HCC) up to 3 months prior to recruitment or will be scheduled for an MRI during the trial period.
* Patient is naïve to any HCC treatment.

Exclusion Criteria:

* Underwent any RFA or TACE or Oral HCC treatments.
* Portal vein thrombosis.
* Prior TIPS placement.
* Severe congestive heart failure (LVEF on echocardiogram < 20%).
* Severe pulmonary hypertension (By echocardiogram, PAS >45 mmHg).
* Uncontrolled diabetes mellitus (HBA1C >9.5%).
* Any autoimmune disorder, which is currently being treated with prednisone or any other immune suppressive medication.
* Previous surgical bypass surgery for morbid obesity (BMI >45).
* Extensive small bowel resection.
* Patients currently receiving total parenteral nutrition if they have contraindications to oral drugs.
* Women who are pregnant or breast feeding.
* Patients with an acute current exacerbation of chronic obstructive pulmonary disease or bronchial asthma.
* Patient has taken drugs that can interfere with octanoate metabolism or can also cause NAFLD independent of the metabolic syndrome, including: corticosteroids, amiodarone, tetracycline, valproic acid, methotrexate, stavudine, zidovudine.
* Patient, based on the opinion of the investigator, should not be enrolled into this study.
* Patient is unable or unwilling to sign informed consent.
* Patients that are participating in other clinical trials evaluating experimental treatments or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morris Sherman, MD, Principal Investigator — Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Suspected HCC: Subjects at high risk for hepatocellular carcinoma (HCC), such as cirrhotics and patients with advanced liver disease will be asked to perform a single Octanoate Breath test, where their breath will be analyzed before and after ingestion of 100 milligrams of Octanoate dissolved in a cup of tap water. The actual breath test procedure lasts approximately one hour.
Period: Overall Study
Arm/Group | Suspected HCC
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Cirrhotic patients with suspected HCC
Arm/Group | Suspected HCC
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Region of Enrollment [Number; unit: participants]
  Israel | 20

OUTCOME MEASURES:

1. Primary Outcome: PDR Peak
Description: PDR peak - the rate at which the 13C labeled substrate is metabolized, percentage dose recovery.
Time Frame: At study day one after one hour
Measure: Mean (Standard Deviation); unit: percentage of dose recovery
Groups:
- Suspected HCC: Subjects at high risk for Hepatocellular carcinoma (HCC), such as cirrhotics and patients with advanced liver disease
Arm/Group | Suspected HCC
Number analyzed (Participants) | 20
percentage of dose recovery | 23.78 (5.51)

ADVERSE EVENTS:
Time Frame: During the one-time Octanoate Breath Test, up to two hours.
Arm/Group | Suspected HCC
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less